CLINICAL TRIAL: NCT06401759
Title: Use of Podcasts in the Education of Hypertension Patients: A Randomized Controlled Study
Brief Title: Use of Podcasts in the Education of Hypertension Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Gülcan Bahçecioğlu Turan, Principal Investigator, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/04-47
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Hypertension
Keywords: Podcast
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Podcast (Experimental)
  Interventions: Behavioral: Podcast
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Podcast — Routine maintenance will be applied.
  Other Names: Control
  Arms: Podcast

SUMMARY:
Hypertension is an important public health problem all over the world due to its high prevalence and its association with increased risk of cardiovascular disease. At the same time, it is a condition in which acquired factors, genetic and metabolic disorders, characterized by increased intra-arterial blood pressure, occur together . According to the World Health Organization, hypertension is defined as systolic blood pressure of 140 mmHg and diastolic blood pressure of 90 mmHg or above According to the Arterial Hypertension Management 2018 Implementation Guide of the European Society of Cardiology and the European Society of Hypertension, it is estimated that there are more than 1 billion hypertension patients in the world and this number will reach 1.5 billion by 2025. In our country, there are approximately 20 million individuals with hypertension. It is thought to be Hypertension treatment is a lifelong process that includes lifestyle changes and patient education along with medical treatment.Turkish Endocrinology and Metabolism.

The aim of hypertension treatment is to ensure that blood pressure decreases to the targeted level, to minimize target organ damage and complications caused by hypertension, to eliminate symptoms and reduce drug side effects, to ensure patient compliance with treatment and to provide self-management skills by enabling the patient to take an active role in his own treatment. The concept of self-management; It includes providing individuals with knowledge and skills regarding disease management, providing support to maintain the individual's self-care, supporting the decision-making process, and helping to recognize and cope with problems. The main goal in hypertension treatment is to control the patient's blood pressure. Achieving and maintaining self-management is also one of the most effective factors in controlling blood pressure. Inadequately treated and low self-management In hypertension patients, blood pressure control is inadequate and health risks increase. Therefore, all strategies implemented to increase self-management in hypertension patients also have positive effects on the individual's blood pressure control and disease prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Education level must be at least primary school level.
* Patients with or without treatment experience
* Being between the ages of 18 and 65
* Being diagnosed with hypertension at least 6 months ago
* Being using at least one hypertensive drug
* Having enough internet to listen to podcasts on Spotify
* Have Spotify supported devices (iOS 14 or above, Android OS 5.0 or above, OS X 10.15 or above, Windows 10 or above)
* Being competent in using a mobile phone
* Having 18.64 points and above in e-health literacy assessment

Exclusion Criteria:

* Those who have physical (speech, hearing impairment, etc.), neurological and psychological problems that prevent them from filling out research forms and participating in training.
* Those who do not have sufficient equipment (mobile phone or computer with internet connection) for podcast training
* Intervention group patients who do not listen to podcasts on Spotify (patients who do not fill out verbally or Google forms (Diary))
* Patients in the control group who were understood to have logged in to their account on Spotify and listened to podcasts.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Hill Bone Hypertension Treatment Compliance Scale | Before and 12 weeks after application
  Measures treatment compliance of hypertension patients. was developed for evaluation. The Cronbach's Alpha value of the scale was found to be between 0.74 and 0.84. The scale is a 4-point Likert type and consists of 14 items and 3 sub-dimensions. The subscales of the scale are Interview (6th, 7th and 8th Questions), Medical (1st, 2nd, 9th, 10th, 11th, 12th, 13th and 14th Questions) and Nutrition (3rd, 14th Questions). 4th and 5th Questions). Question 6 on the scale is reverse coded. The total score range on the scale varies between 0 and 42. If the person gives the most positive answers to all questions and receives a total of 0 points, he or she is considered fully compliant. Scores outside zero indicate the degree of non-compliance. Since the questions are in the negative type of questions, the compliance decreases as the score increases.
Self-Care Management Scale in Chronic Diseases | Before and 12 weeks after application
  It was developed to evaluate self-care management in chronic diseases. (The scale has a 5-point Likert structure (1=strongly disagree, 2=disagree, 3=undecided, 4=agree, 5=strongly agree) and consists of 35 items. The scale consists of two sub-dimensions. These sub-dimensions are: "self-protection" ( articles 2, 6, 8, 11, 15, 18, 19, 20, 22, 23, 25-34), and "social protection" (articles 1, 3, 4, 5, 7, 9, 10, 12, 13 , 14, 16, 17, 21, 24 and 35 items. The 3rd, 15th, 19th and 28th items in the scale are negative expressions. The total scores that can be obtained from the scale vary between 35 and 175 points. It indicates that the individual's self-care management also increases

CONTACTS AND LOCATIONS:
Locations (1):
- Fırat university, Elâzığ, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
after the project is finished